CLINICAL TRIAL: NCT01565486
Title: Comparison of Surgical Outcomes Between Papillary Thyroid Cancer Patients Treated With the Harmonic ACE® Scalpel and LigaSure Precise™ Instrument During Conventional Thyroidectomy: A Single-blind Prospective Randomized Controlled Trial
Brief Title: Safety and Efficacy Study of Ultrasonic Coagulation Device and Bipolar Energy Sealing System
Acronym: UCBEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Ja Seong Bae, MD, phD, Division of Breast and Endocrine Surgery, Department of Surgery, The Catholic University of Korea College of Medicine, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC11DISI0534
Record Dates: First submitted 2011-09-02; First posted 2012-03-28 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Thyroid Cancer
Keywords: operation time; complication rate; costs; admission time; RFS; OS
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasonic coagulation device (Other): Comparison of Surgical Outcomes Between Papillary Thyroid Cancer Patients Treated with the Ultrasonic coagulation device (Harmonic ACE® Scalpel) and the bipolar energy sealing system (LigaSure Precise) during Conventional Thyroidectomy
  Interventions: Device: Ultrasonic coagulation device (Harmonic ACE® scalpel)
- Bipolar Energy Sealing System (Other): Comparison of Surgical Outcomes Between Papillary Thyroid Cancer Patients Treated with the Ultrasonic coagulation device (Harmonic ACE® Scalpel) and the bipolar energy sealing system (LigaSure Precise) during Conventional Thyroidectomy
  Interventions: Device: bipolar energy sealing system (LigaSure Precise)

INTERVENTIONS:
Device: Ultrasonic coagulation device (Harmonic ACE® scalpel) — Comparison of Surgical Outcomes Between Papillary Thyroid Cancer Patients Treated with the Ultrasonic coagulation device (Harmonic ACE® Scalpel) and the bipolar energy sealing system (LigaSure Precise) during Conventional Thyroidectomy
  Other Names: Harmonic ACE® scalpel
  Arms: Ultrasonic coagulation device
Device: bipolar energy sealing system (LigaSure Precise) — Comparison of Surgical Outcomes Between Papillary Thyroid Cancer Patients Treated with the Ultrasonic coagulation device (Harmonic ACE® Scalpel) and the bipolar energy sealing system (LigaSure Precise) during Conventional Thyroidectomy
  Other Names: LigaSure Precise instrument
  Arms: Bipolar Energy Sealing System

SUMMARY:
The aim of the study is to evaluate differences between use of Ultrasonic Coagulation Device (New Harmonic ACE™, Ethicon endo-surgery) and Bipolar Energy Sealing System (LigaSure Precise™, Covidien) in surgery for thyroid cancer.

Abbreviations: Ultrasonic Coagulation Device (UC), Bipolar Energy Sealing System (BES), Recurrence-free survival (RFS), Overall survival (OS)

DETAILED DESCRIPTION:
Background: Thyroid is an organ that has abundant vessels. In thyroid surgery, it should be cautious to avoid injury of the recurrent laryngeal nerve and parathyroid, thus careful hemostasis during surgery is crucial for surgeons who perform thyroid surgery. Recently, there have been significant advances in vessel sealing systems for the occlusion of vessels during surgery as endoscopic surgery has been developed. UC and BES are now commonly used in thyroid surgery. However, only a few studies have compared the two surgical devices to determine which technique is superior in terms of operative time and complication rate. Thus, this single-blind prospective randomized trial is conducted to determine if there was a difference in operative time, complication rate, postoperative drainage volume, admission time, cost, and, furthermore, oncologic outcomes (RFS and OS) between the two surgical devices in surgery for thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

1. an age between 20 and 80 years old who are diagnosed as thyroid cancer or suspicious papillary thyroid cancer in fine needle aspiration biopsy
2. patients who are agree with the study enrollment

Exclusion Criteria:

1. an age under 20 or over 80 years
2. severe co-morbidities that were contraindications for thyroid surgery (e.g., severe liver, heart, kidney, or pulmonary problems)
3. a lack of consent to participate in the study
4. the inability to include a patient in clinical trials according to the regulations or laws in Korea
5. the inability to complete regular follow-up visits (e.g., immigration)
6. the use of modified radical neck dissection due to lateral neck node metastasis
7. prior thyroid surgery or cervical irradiation
8. active enrollment in another clinical trial
9. the intention of the patient to undergo an additional operation at the time of the thyroid surgery (e.g., mastectomy and thyroidectomy at the same time)
10. the desire to undergo endoscopic or robot-assisted thyroidectomy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
operation time | from skin incision to skin closure at an average time of 60 min to 160 min according to the extent of surgery
  from skin incision to skin closure

SECONDARY OUTCOMES:
postoperative complications | at 3 hours, 1, 2, 3, 10 days and 1 months after surgery and 6 months and every 1 years after surgery
postoperative drainage volume | estimated until the drain tube is removed at the average of 4 to 7 days according to the extent of surgery
admission time | documented when the patient leaves the hospital at an average time of 5 to 10 days according to the extent of surgery
Cost | documented when the patient leaves the hospital at an average time of 5 to 10 days according to the extent of surgery
Relapse-free survival (RFS) | from date of surgery until date of first documented recurrence or date of death from any cause, whichever came first, accessed up to 60 months
Overall Survival (OS) | from date of surgery until date of death from any cause, accessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Ja Seong Bae, MD,phD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seocho-gu, Seoul, South Korea